CLINICAL TRIAL: NCT04860141
Title: Efficacy of Preoperative Administration of Gabapentin in Managing Intraoperative and Postoperative Pain From Third Molar Extractions.
Brief Title: Efficacy of Preoperative Administration of Gabapentin in 3rd Molar Dental Extraction.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5200474
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dental Pain and Sensation Disorder; Pain, Postoperative
Keywords: gabapentin; third molar extraction; postoperative pain; intraoperative pain; opioid reduction; narcotic reduction
MeSH Terms: conditions — Toothache; Sensation Disorders; Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: * Only the allocator knows the computer generated randomization scheme and this will be strictly controlled. The allocator will not be directly involved in the patient care.
  * The allocator will also pre-package a pill in a small bag so that a distributor does not know which medication is being given to the patient.
  * Gabapentin and placebo pills will be formulated by an investigational pharmacist to ensure both pills are identical in shape and form to further reduce bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gabapentin group (Experimental): The patient in this group will take gabapentin 600mg PO 2 hours prior to his or her surgery.
  Interventions: Drug: Gabapentin 600mg
- Placebo group (Placebo Comparator): The patient in this group will take a placebo that looks like gabapentin PO 2 hours prior to his or her surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin 600mg — The patient will take gabapentin 600mg 2 hours prior to the procedure
  Arms: Gabapentin group
Drug: Placebo — the patient will take a pill that looks like gabapentin 2 hours prior to the procedure
  Arms: Placebo group

SUMMARY:
This study is a double-blind, randomized, prospective, placebo-controlled single-center clinical research study in which 600 mg of gabapentin or placebo will be administered 2 hours preoperatively to 49 patients each undergoing wisdom teeth extraction. We will measure intraoperative opioid use, severity of pain, the number of analgesics taken, and side effect profiles (e.g. nausea/vomiting, dizziness) at the following intervals, 4 hour, 8 hour, 12 hour, 24, and 72 hour post-procedure.

DETAILED DESCRIPTION:
Since the 1990s, the amount of prescribed opioids has begun growing. According to the Center for Disease Control, more than 130 people die every day due to opioid overdose. Many medical and surgical specialities have devised various methods to decrease opioid use with adequate pain control. One notable method is preoperative administration of gabapentin. Gabapentin, a prescribed medication, is an anticonvulsant medication used to treat partial seizures, neuropathic pain (e.g.

diabetic neuropathy, postherpetic neuralgia, and central neuropathic pain), hot flashes, and restless legs syndrome . Various surgical specialties such as otolaryngology, plastics, general surgery, obstetrics/gynecology have tested the efficacy of gabapentin in reducing postoperative opioid usage without compromising pain control and the result is promising. However, this study has not been done in oral and maxillofacial surgery. The objectives of the study is to determine if preoperative administration of gabapentin can decrease intraoperative and postoperative use of opioid and provide adequate pain control when used with non-opioid pain regimen.

On the day of consultation visit, subjects will be screened and evaluated by oral and maxillofacial surgery residents. Those who meet the inclusion criteria will be enrolled in the study. They will then be randomly divided into following groups:

* Group 1a: 49 subjects undergoing wisdom teeth extraction will be receiving 600mg gabapentin PO preoperatively
* Group 1b: 49 subjects undergoing wisdom teeth extraction will be receiving placebo PO preoperatively.

A subject then will be given a small bag that contains either a gabapentin pill or a placebo pill depending on which group that he or she is assigned to. The subject will be asked to take 600mg of gabapentin or a placebo pill 2 hours prior to their procedure (vs. current standard of care is no pre-medication). On the day of the procedure, they will be accompanied by a guardian or a family member to the clinic. The Procedure will be done by a senior or a chief level resident with supervision of an attending surgeon. Intraoperative opioid use will be recorded on a standardized anesthesia sheet. All cases will include IV sedation that involves a concoction of fentanyl, midazolam, propofol, ketamine, and dexamethasone. The medications will be given in boluses depending on their weight but not necessarily strictly kg-based. For example, fentanyl will be given between 25 -50mcg, midazolam 2.5-5mg, propofol 10-40mg and ketamine 10-50mg. Local anesthesia with 2% lidocaine with 1:100,000 epinephrine will also be given after sedation. Additional doses of local anesthetic can be given if the patient experiences sharp pain. Additional doses of propofol and/or fentanyl can be given if the patient's systolic blood pressure increases by 10 mmHg or heart rate increases by 20 bpm acutely. All used anesthetics will be recorded. After the procedure, standard postoperative pain regimen will be prescribed including 28 tablets of ibuprofen 600mg PO q6h prn pain and 12 tablets of Norco 5/325mg PO q6h prn pain with an instruction to take Norco only when a subject is in severe pain (pain level greater than 7 out of 10). To assess the severity of pain and its impact on functioning, scientists developed Brief Pain Inventory from which Modified Brief pain inventory (MBPI) was created to better fit the need for our research; MBPI will not only ask the severity of pain but also the number of analgesics taken and side effect profiles (e.g. nausea/vomiting, dizziness) at the following intervals, 4 hour, 8 hour, 12 hour, 24, and 72 hour post-procedure. The patient is to turn in the MBPI form during their 1 week postoperative follow up visit. If for any reason, the patient misses the follow up appointment, we will try to reschedule their visit within 5 days. If the patient does not show up at all, our members will find out the reason for the no show and record it for the publication purpose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at or older than 18.
* Screened body mass index (BMI) between 18-35 kg/m2.
* American Society of Anesthesiologists Classification I and II.
* Subjects must be willing and able to comply with protocol requirements.
* Subjects must be able to understand the informed consent and must be able to sign a written informed consent form prior to the initiation of any study procedures.
* A subject must have at least 1 partial or fully impacted third molar tooth removal.

Exclusion Criteria:

* hypersensitivity to gabapentinoids;
* history of chronic opioid or gabapentin usage (regular use of opioids >3 months)
* history of recreational drug usage
* a history or clinical manifestations of significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, musculoskeletal, psychiatric, or immunologic disorder, any acute, clinically significant illness or condition within 14 days prior to Day 1.
* Patients with baseline pain.
* Patients with any oral pathology will be excluded.
* Pregnant or breastfeeding patients
* An individual not legally competent to consent (e.g., incapacitated individuals, incompetents, minors)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
opioid use | 4 hour postoperatively
  assess the number of opioid pills (norco 5/325mg) taken postoperatively. #of pills that a patient takes.
opioid use | 8 hour postoperatively
  assess the number of opioid pills (norco 5/325mg) taken postoperatively. #of pills that a patient takes.
opioid use | 12 hour postoperatively
  assess the number of opioid pills (norco 5/325mg) taken postoperatively. #of pills that a patient takes.
opioid use | 48 hour postoperatively
  assess the number of opioid pills (norco 5/325mg) taken postoperatively. #of pills that a patient takes.
opioid use | 72 hour postoperatively
  assess the number of opioid pills (norco 5/325mg) taken postoperatively. #of pills that a patient takes.
intraoperative fentanyl use | during the surgical procedure
  assess amount of fentanyl given intraoperatively. mcg of fentanyl given in a case.

SECONDARY OUTCOMES:
pain control | 4 hour postoperatively
  assess amount of pain that the patient is in by using modified brief pain index. (0 is no pain at all, 10 is the worst pain- interfering with one's everyday activity)
pain control | 8 hour postoperatively
  assess amount of pain that the patient is in by using modified brief pain index. (0 is no pain at all, 10 is the worst pain- interfering with one's everyday activity)
pain control | 12 hour postoperatively
  assess amount of pain that the patient is in by using modified brief pain index (0 is no pain at all, 10 is the worst pain- interfering with one's everyday activity)
pain control | 24 hour postoperatively
  assess amount of pain that the patient is in by using modified brief pain index (0 is no pain at all, 10 is the worst pain- interfering with one's everyday activity)
pain control | 48 hour postoperatively
  assess amount of pain that the patient is in by using modified brief pain index (0 is no pain at all, 10 is the worst pain- interfering with one's everyday activity)
pain control | 72 hour postoperatively
  assess amount of pain that the patient is in by using modified brief pain index (0 is no pain at all, 10 is the worst pain- interfering with one's everyday activity)
nausea | within 72 hour postoperatively
  If the pt is having nausea any time within 72hrs. Yes or No.
Vomiting | within 72 hour postoperatively
  If the pt is having vomiting any time within 72hrs. Yes or No.
Dizziness | within 72 hour postoperatively
  If the pt is having dizziness any time within 72hrs. Yes or No.
Drowsiness | within 72 hour postoperatively
  If the pt is having drowsiness any time within 72hrs. Yes or No.
pain interfering in general activity | within 72 hours postoperatively
  0 is not interference at all, 10 is severely interfering with life.
pain interfering in mood | within 72 hours postoperatively
  pain interfering in mood; 0 is not interference at all, 10 is severely interfering with life.
pain interfering in normal work | within 72 hours postoperatively
  pain interfering in normal work; 0 is not interference at all, 10 is severely interfering with life.
pain interfering in relations with other people | within 72 hours postoperatively
  pain interfering in relations with other people; 0 is not interference at all, 10 is severely interfering with life.
pain interfering in sleep | within 72 hours postoperatively
  pain interfering in sleep; 0 is not interference at all, 10 is severely interfering with life.
pain interfering in enjoyment in life | within 72 hours postoperatively
  pain interfering in enjoyment in life; 0 is not interference at all, 10 is severely interfering with life.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Viet, DDS MD PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
As of right now we do not intend to share any study protocol or statistical analysis plan other than what will be described in the published documentation.

REFERENCES:
- [Background] Turan A, Memis D, Karamanlioglu B, Yagiz R, Pamukcu Z, Yavuz E. The analgesic effects of gabapentin in monitored anesthesia care for ear-nose-throat surgery. Anesth Analg. 2004 Aug;99(2):375-8, table of contents. doi: 10.1213/01.ANE.0000136646.11737.7B. PMID 15271709
- [Background] Salama ER, Amer AF. The effect of pre-emptive gabapentin on anaesthetic and analgesic requirements in patients undergoing rhinoplasty: A prospective randomised study. Indian J Anaesth. 2018 Mar;62(3):197-201. doi: 10.4103/ija.IJA_736_17. PMID 29643553
- [Background] Han C, Li XD, Jiang HQ, Ma JX, Ma XL. The use of gabapentin in the management of postoperative pain after total knee arthroplasty: A PRISMA-compliant meta-analysis of randomized controlled trials. Medicine (Baltimore). 2016 Jun;95(23):e3883. doi: 10.1097/MD.0000000000003883. PMID 27281103
- [Background] Grover VK, Mathew PJ, Yaddanapudi S, Sehgal S. A single dose of preoperative gabapentin for pain reduction and requirement of morphine after total mastectomy and axillary dissection: randomized placebo-controlled double-blind trial. J Postgrad Med. 2009 Oct-Dec;55(4):257-60. doi: 10.4103/0022-3859.58928. PMID 20083871
- [Background] Crisologo PA, Monson EK, Atway SA. Gabapentin as an Adjunct to Standard Postoperative Pain Management Protocol in Lower Extremity Surgery. J Foot Ankle Surg. 2018 Jul-Aug;57(4):781-784. doi: 10.1053/j.jfas.2018.02.005. Epub 2018 May 7. PMID 29748103
- [Background] Felder L, Saccone G, Scuotto S, Monks DT, Carvalho JCA, Zullo F, Berghella V. Perioperative gabapentin and post cesarean pain control: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2019 Feb;233:98-106. doi: 10.1016/j.ejogrb.2018.11.026. Epub 2018 Dec 12. PMID 30583095
- [Background] Quintero GC. Review about gabapentin misuse, interactions, contraindications and side effects. J Exp Pharmacol. 2017 Feb 9;9:13-21. doi: 10.2147/JEP.S124391. eCollection 2017. PMID 28223849
- [Background] Sanders JG, Dawes PJ. Gabapentin for Perioperative Analgesia in Otorhinolaryngology-Head and Neck Surgery: Systematic Review. Otolaryngol Head Neck Surg. 2016 Dec;155(6):893-903. doi: 10.1177/0194599816659042. Epub 2016 Jul 26. PMID 27459955